CLINICAL TRIAL: NCT06662240
Title: Effect of Vibration Anesthesia on Pain, Ecchymosis and Comfort Level in Subcutaneous Heparin Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Meltem SIRIN GOK, assistant professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15653993494; TYL-2023-12968 (Other Grant/Funding Number: Scientific Research Projects (BAP) Coordination Unit under the Rectorate of Atatürk University)
Record Dates: First submitted 2024-08-06; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Pain; Ecchymosis; Comfort
Keywords: pain; ecchymosis; comfort; vibration anesthesia; subcutaneous injection; nursing; heparin
MeSH Terms: conditions — Pain; Ecchymosis

STUDY DESIGN:
Intervention Model Description: Each patient in the experimental and control groups received two subcutaneous injections. Each patient in the experimental group received one injection with vibration and one without vibration. Each patient in the control group received two injections without vibration. The purpose of administering two injections was to obtain control data within the experimental group by controlling individual factors related to the dependent variables of the study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Application of vibration anesthesia (Experimental): In addition to the routine injection protocol performed from the abdominal region, the vibration device was kept on the injection site by the investigator for 3 minutes just before the injection, the vibration device was removed from the injection site, and the injection was performed by the investigator immediately afterwards.
  Interventions: Device: The effect of vibration anesthesia on pain, ecchymosis and comfort level in subcutaneous heparin injection
- Subcutaneous Heparin Injection without Vibration Anesthesia (Standard) (No Intervention): The patient will be informed about the procedure and consent will be obtained. Hands will be washed before the procedure and the abdomen, excluding the 5 cm2 area around the umbilicus, will be used for abdominal SC injection.
  During abdominal SC injections, the patient will be given a semi-fowler position that will be comfortable and does not complicate the injection, and the injection site will be cleaned with 70% alcohol cotton wool with circular movements from the center to the outside and left to dry.
  After the area dries, the skin and subcutaneous tissue in the injection area will be grasped between the thumb and index fingers.
  For injections, a 25 gauge, 1.26 cm needle length, air-locked, ready-to-use syringe containing DMAH (enoxaparin sodium) will be used to enter the tissue at a 90° angle, not aspiration will be performed, the drug will be applied for 10 seconds and the drug will be exited at a 90° angle.

INTERVENTIONS:
Device: The effect of vibration anesthesia on pain, ecchymosis and comfort level in subcutaneous heparin injection — The patient in the experimental group received one vibrating injection and one non-vibrating injection into the abdomen. The patient in the control group received 2 standard subcutaneous injections in the abdomen without vibration.
  Arms: Application of vibration anesthesia

SUMMARY:
The aim of this study is to determine the effect of vibration anesthesia on injection pain, ecchymosis and comfort level in subcutaneous heparin injection.This study was conducted in a randomized controlled experimental design.

DETAILED DESCRIPTION:
Population and Sample of the Research

The population of the research consisted of the doses administered by subcutaneous heparin injection in the chest diseases clinic of Atatürk University Health Research and Application Center. Among the total data related to the study, 162 patients were evaluated. There were 28 patients who met the study eligibility criteria and 18 who refused to participate in its terms. 116 patients who volunteered to comply with the data collection, total fee criteria and participate will be assigned to the experimental group, 58 patients to the control group, and 58 patients to the control group by randomization. 8 patients from the experimental group left the study because they were discharged early. In the control group, 6 patients were discharged early rather than 2 patients in the study. Training data was completed with 50 patients in both experimental and control classes. To determine whether the sample size was sufficient, post-hoc power analysis was calculated with the G*Power 3.1.9.7 program.

Post hoc power analysis of the study was determined to be over 0.90 with a margin of error of 0.05 for the analysis conducted on the basis of t test in independent groups of the 2nd combination application. Completed with 50 patients in both the experimental and control groups. Post-hoc power analysis was calculated with the G*Power 3.1.9.7 program to determine whether the sample size was sufficient. The power of the study was determined to be above 0.90 with a margin of error of 0.05 for the post hoc power analysis based on the t test in independent groups for the 2nd injection application.

Inclusion Criteria

* Clexane (Enoxaparin Sodium) 0.6 ml SC 1x1 DMAH treatment (0.6 ml heparin was preferred because pain and ecchymosis may be less at a dose of 0.4 ml heparin and the incidence of pain and ecchymosis may increase at a dose of 0.8 ml Clexane.
* No cognitive, physical or mental impairment that prevented them from answering the questions,
* 18 years of age or older,
* No previous known coagulation disorders,
* Platelet value between 150,000 and 300,000/millimeter cubed,
* PTZ value between 10-14 seconds,
* aPTT value between 20-40 seconds,
* INR value between 0.8-1.2,
* No incision, infection, ecchymosis, hematoma, scar tissue in the abdominal region
* No needle phobia
* Not taking pain medication in the last 12 hours
* No abdominal pain
* No other invasive procedures in the abdominal region
* SC heparin not administered by subcutaneous, intramuscular or intradermal injection,
* Patients with no known allergy to heparin,
* Patients with a body mass index above 18.5 were included in the study.

Non-reception Criteria

* Uncommunicative,
* Have any disease that may cause sensory loss (diabetic neuropathy, stroke, multiple sclerosis, etc.),
* Receiving hemodialysis,
* Patients with a history of pregnancy were excluded from the study.

Exclusion Criteria

* The patient wishes to withdraw from the study,
* Discharge of the patient within 48 hours after inclusion in the study,
* Change of the patient's clexan dose
* Another injection in the abdomen during the study.

Data Collection Tools:

The data of the study will be collected using 4 forms. Patient Introduction Form, Octoberosis Measurement Tool, Visual Analog Scale, Visual Analog Comfort Scale, Patient Follow-up Form will be used.

Patient Introduction Form It is a form prepared in line with the literature that includes the information of the patients (gender, age, marital status, educational status, employment status, body mass index, chronic disease, continuous medication use, smoking status).

Ecchymosis Measurement Tool A transparent measuring tool was used to measure the ecchymosis at the injection site. The transparent measuring tool was placed on the ecchymosis and the borders of the ecchymosis were drawn with an acetate pen; then, the size of the ecchymosis was determined in mm2 by placing the transparent measuring tool on a millimeter measuring paper and recorded on the patient follow-up form. The size of the ecchymosis was measured at 48 hours after injection. It is reported that ecchymosis after subcutaneous heparin injection is most prominent after 48 hours . Based on the literature, discoloration smaller than 2 mm2 was considered as "no ecchymosis", and the size of discoloration of 2 mm2 or more was measured.

Visual Analog Pain Scale The Visual Analog Scale (VAS) is a scale system used to convert some characteristics that cannot be quantitatively measured into numerical values. VAS pain was used to measure the intensity of pain during injection. The VAS pain scale is expressed as "0=No pain, 10=Unbearable pain" on a 10 cm horizontal line. Patients were asked to mark the intensity of pain experienced during subcutaneous injection with an X on the scale. It is a widely used valid scale.

Visual Analog Comfort Scale The VAS comfort is a 10 cm long horizontal measurement tool that starts with "most comfortable" and ends with "most uncomfortable". Patients rated their comfort level with this scale. For a better understanding of the term comfort by patients, they were asked to indicate their "comfort, satisfaction or level of comfort with the injection" on the scale. It is a valid scale widely used to assess comfort.

Patient Follow-up Form The patient follow-up form records the date and time of the injection, the patient's name or pseudonym, the group to which the patient belongs, the standard injection method with or without vibration, the injection site, pain intensity, comfort level and ecchymosis size.

Vibration Anesthesia Device The vibration anesthesia device is a reusable, handheld device with a battery-powered motor and a vibration frequency of approximately 6000 times per minute. Based on the Gate Control Theory, one of the pain theories, vibration anesthesia is used to reduce pain in injections . The vibration anesthesia device helps to close the pain gate by stimulating large diameter nerve fibers during the application. By producing low-frequency vibrations, the device affects the nerves under the skin and prevents pain signals from reaching the brain.

Standard Subcutaneous Heparin Injection without Vibration The steps of injection are given below.

1. Materials were prepared. Drug order was checked.
2. Hand hygiene was ensured. The identity of the patient was verified.
3. The door of the room was closed and the patient's privacy was ensured.
4. The patient was informed about the research. Informed written consent was obtained.
5. Disposable gloves were worn. The lower abdominal area outside the 5 cm2 area around the navel was used for injection.
6. The patient was given a semifowler position to relax the abdominal region. The injection site was gently cleaned with 70% alcohol cotton wool in a 5 cm wide circular motion from the center to the outside and allowed to dry.
7. After the area had dried, the skin and subcutaneous tissue at the injection site was grasped or held between the thumb and index fingers according to the patient's weight.
8. Ready-to-use syringes with 25 gauge, 1.26 cm needle length, airlock, and DMAH enoxaparin sodium were used for injection.
9. The needle was serially inserted into the tissue at an angle of 45-90° according to the patient's body mass index. The skin was left free. After insertion, no aspiration was performed for blood control.
10. The drug was injected for 10 seconds/ml. The needle was removed serially at the same angle by applying dry cotton over the injection site without pressing.
11. After the needle was removed, pressure was applied with dry cotton for 10 seconds. To standardize the applied pressure, the whitening of the nail tip of the finger applying pressure was accepted as a criterion . No massage was performed.
12. The injection site was circled with an acetate pen (8 cm around the injection site).
13. The patient was informed not to scratch, wash or rub the injection site. In addition, both the patient and the clinic nurse were informed not to perform subcutaneous injection or any application to the abdominal region until ecchymosis was evaluated at the injection site.
14. Immediately after the injection, pain intensity was measured and comfort levels were evaluated as specified in the patient follow-up form, and ecchymosis size was measured at 48 hours after the injection.
15. The materials used were separated in accordance with medical waste rules.
16. The patient was given a comfortable position.
17. Gloves were removed and hand hygiene was ensured.

Vibratory Subcutaneous Heparin Injection Steps 1-6 were performed as in standard subcutaneous heparin injection without vibration. The vibration anesthesia device was wiped with 70% alcohol cotton wool and allowed to dry. The researcher held the vibration anesthesia device for 3 minutes on the exact injection point just before the injection. Immediately afterwards, the skin and subcutaneous tissue were grasped and subcutaneous injection was performed according to steps 7-17 of the standard subcutaneous heparin injection.

Data Collection Patients were informed about the study and their consent was obtained. Before the injection, the patients were informed that they would be asked about the severity of pain they felt after the injection and their comfort level. Platelet, PTZ, aPTT, aPTT, INR values determined in the last 24 hours were checked. The abdomen was chosen as the injection site in the study. Since muscle movements are less in the abdomen, patient-specific differences may be less in the follow-up of ecchymosis after injection compared to the arm and leg. Another reason for choosing the abdominal region is that clinical nurses mostly prefer the arm and leg regions for heparin injections outside the study. The abdominal region of the patient was evaluated for incision, infection, ecchymosis and/or hematoma, and scar tissue. All injections in the experimental and control groups were performed by the same investigator. Patients and clinic nurses were informed not to perform another injection in the injection site and not to wash the injection site for 48 hours for ecchymosis follow-up.

Experimental Group The patients in the experimental group were administered subcutaneous heparin injections with and without vibration, the order of which was determined by lottery, at one day intervals. The purpose of administering two injections with and without vibration to the experimental group was to obtain control data within the experimental group by controlling individual factors related to the dependent variables of the study. The non-vibrated injection was performed according to the standard subcutaneous heparin injection steps. For vibratory injection, vibration anesthesia was applied to the injection site for three minutes just before the procedure , followed by standard injection steps. The right and left sides of the lower abdomen were randomly used as the injection site. The injection site was circled with an acetate pen.

Control Group In the control group, two non-vibrated SC heparin injections were administered 24 hours apart. The aim of administering two non-vibrated injections to the control group was to obtain control data within the control group by controlling individual factors related to the dependent variables of the study. In the control group, injections were performed according to the steps of standard subcutaneous heparin injection without vibration. The right and left sides of the lower abdomen were randomly used as the injection site. The injection site was circled with an acetate pen.

Randomization Randomization was performed in a computerized environment using the website https://www.randomizer.org/web. In randomization, each patient was assigned to only one group with a 1:1 chance of selection. Randomization was performed by a statistical expert who was not involved in the research process. According to the randomization outputs, patients' numbers were listed in two groups. The lottery method was used to determine the two groups as experimental and control groups. The first group drawn first was assigned to the experimental group and the second group drawn second was assigned to the control group. Patients who met the inclusion criteria were numbered according to the order of hospitalization. Patients were identified as being in the experimental or control group according to their numbers.

The order of the non-vibratory and vibratory standard injections administered to the patients in the experimental group was determined randomly by lottery method. Injection methods were coded as A and B. The researcher wrote the names of the injection methods on two pieces of paper and drew lots to determine which injection would be coded A and B. The first method drawn was vibratory injection: A and the second method drawn was non-vibratory injection: B. The injection order was classified as AB, BA. Then, for each patient, which of the AB or BA injection order would be chosen was determined by lottery.

Another method used to prevent bias in experimental studies is blinding. The main purpose of blinding is to obtain and evaluate the results objectively. Patients were not informed that they were in the experimental or control group. Patients were blind to the hypotheses of the study. During the data analysis phase, the experimental group was coded as A and the control group as B, and the statistician was blinded to the study.

This randomized controlled experimental study was conducted according to "The CONSORT-Outcomes 2022 Extension guidelines.

Data Evaluation Data were analyzed with the SPSS for Windows 22 software package . Continuous data were presented as mean ± standard deviation and categorical data were presented as frequency and percentage. Chi-square test was used to compare categorical demographic data between groups. Kurtosis and skewness values in the range of ±2 indicate that continuous variables are normally distributed . It was determined that ecchymosis size was not normally distributed in the experimental and control groups, while other variables were normally distributed. In intergroup comparison, independent samples t test was performed for normally distributed parameters and Mann Whitney U analysis was performed for non-normally distributed measurements. In intragroup comparison, paired sample t test was used for normally distributed parameters and Wilcoxon sign test was used for non-normally distributed parameters. In the study, p<0.05 was considered statistically significant. The effect size of the difference was calculated if a difference was found in intra- and inter-group comparisons. The effect size was classified as insignificant (0.0-0.19), low (0.20-0.49), moderate (0.50-0.79) and high effect (≥0.80).

Financial Source This research was supported by the Scientific Research Projects (BAP) Coordination Unit of Atatürk University Rectorate as project number TYL-2023-12968.

ELIGIBILITY:
Inclusion Criteria

* Clexane (Enoxaparin Sodium) 0.6 ml SC 1x1 DMAH treatment (0.6 ml heparin was preferred because pain and ecchymosis may be less at a dose of 0.4 ml heparin and the incidence of pain and ecchymosis may increase at a dose of 0.8 ml Clexane .
* No cognitive, physical or mental impairment that prevented them from answering the questions,
* 18 years of age or older,
* No previous known coagulation disorders,
* Platelet value between 150,000 and 300,000/millimeter cubed,
* PTZ value between 10-14 seconds,
* aPTT value between 20-40 seconds,
* INR value between 0.8-1.2,
* No incision, infection, ecchymosis, hematoma, scar tissue in the abdominal region
* No needle phobia
* Not taking pain medication in the last 12 hours
* No abdominal pain
* No other invasive procedures in the abdominal region
* SC heparin not administered by subcutaneous, intramuscular or intradermal injection,
* Patients with no known allergy to heparin,
* Patients with a body mass index above 18.5 were included in the study.

Non-reception Criteria

* Uncommunicative,
* Have any disease that may cause sensory loss (diabetic neuropathy, stroke, multiple sclerosis, etc.),
* Receiving hemodialysis,
* Patients with a history of pregnancy were excluded from the study.

Exclusion Criteria

-The patient follow-up form records the date and time of the injection, the patient's name or pseudonym, the group to which the patient belongs, the standard injection method with or without vibration, the injection site, pain intensity, comfort level and ecchymosis size.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Ecchymosis Measurement Tool | 7 months
  A transparent measuring tool was used to measure the ecchymosis at the injection site. The transparent measuring tool was placed on the ecchymosis and the borders of the ecchymosis were drawn with an acetate pen; then, the size of the ecchymosis was determined in mm2 by placing the transparent measuring tool on a millimeter measuring paper and recorded on the patient follow-up form. The size of the ecchymosis was measured at 48 hours after injection. It is reported that ecchymosis after subcutaneous heparin injection is most prominent after 48 hours. Based on the literature, discoloration smaller than 2 mm2 was considered as "no ecchymosis", and the size of discoloration of 2 mm2 or more was measured.
Patient Introduction Form | 7 months
  It is a form prepared in line with the literature that includes the information of the patients (gender, age, marital status, educational status, employment status, body mass index, chronic disease, continuous medication use, smoking status).
Visual Analog Pain Scale | 7 months
  The Visual Analog Scale (VAS) is a scale system used to convert some characteristics that cannot be quantitatively measured into numerical values. VAS pain was used to measure the intensity of pain during injection. The VAS pain scale is expressed as "0=No pain, 10=Unbearable pain" on a 10 cm horizontal line. Patients were asked to mark the intensity of pain experienced during subcutaneous injection with an X on the scale. It is a widely used valid scale.
Visual Analog Comfort Scale | 7 months
  The VAS comfort is a 10 cm long horizontal measurement tool that starts with "most comfortable" and ends with "most uncomfortable". Patients rated their comfort level with this scale. For a better understanding of the term comfort by patients, they were asked to indicate their "comfort, satisfaction or level of comfort with the injection" on the scale. It is a valid scale widely used to assess comfort.
Patient Follow-up Form | 7 months
  The patient follow-up form records the date and time of the injection, the patient's name or pseudonym, the group to which the patient belongs, the standard injection method with or without vibration, the injection site, pain intensity, comfort level and ecchymosis size.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem SIRIN GOK, Assistant Professor, Study Director — meltemsirin@atauni.edu.tr; Yaprak BAGA, Research Assistant, Principal Investigator — yaprak.baga@atauni.edu.tr
Locations (1):
- Meltem, Erzurum, yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No